CLINICAL TRIAL: NCT00835458
Title: Closure of Fistulas and Perforations Endoscopically to Avoid Laparoscopic or Open Surgery
Brief Title: Endoscopic Treatment of Intestinal Fistulas and Perforations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Legacy Health System (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Lee Swanstrom, Legacy Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS GRANT#25206
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Fistula
Keywords: gastric fistula; perforation; endoscopy; closure; endolumenal
MeSH Terms: conditions — Gastric Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: gastro-gastric fistula closure — The mucosa surrounding the orifice of the fistula will be ablated using standard endoscopic techniques. Remnants of mucosa will be treated with argon-plasma coagulation. The mucosa free orifice of the fistula will be closed using the Tissue Apposition System. Tissue anchors with attached threads will be deployed through the intestinal wall full thickness using delivery needles through the working channel of the endoscope. After two anchors are deployed on both sides of the fistulas' orifice a knotting element will be cinched down to approximate the two sides of the fistulas' orifice. The procedure will be repeated until the fistulas' orifice is securely closed.
  Other Names: Tissue Apposition System; TAS; 510(k) approval # K070151

SUMMARY:
Background: T-shaped tissue anchors have promise to close incisions and perforations of the intestines securely. The closure of perforations, gastro-gastric, or intestinal fistulas usually requires invasive open or laparoscopic surgery under general anesthesia and can be complex surgeries due to their reoperative or inflammatory nature.

Objective: The proposed use of full thickness tissue anchors adds a new surgical aspect to the endoscopic treatment of fistulas and perforations by offering a robust suture like closure of defects. Instead of a 20 cm abdominal incision or 3 or 4 one centimeter incisions with the related postoperative morbidity an endoscopic technique is used which requires no postoperative limitation of activities.

Methods: In this study the investigators propose to use an endoscopic technique that eliminates the need for open or laparoscopic surgery and provides a more robust endoscopic repair than is possible with traditional endoscopic tools. Patients who are scheduled to undergo surgery for intestinal fistulas will be screened for study eligibility. Patients who are scheduled to undergo complex polypectomy, or submucosal dissection will be screened for study eligibility and informed about all possible therapies in case of an iatrogenic perforation (open - laparoscopic surgery, endoscopic clipping, endoscopic closure with tissue anchors). A commercially available flexible endoscope will be inserted through the mouth and the fistula or perforation will be closed using the Tissue Approximation System (Ethicon Endo Surgery, Cincinnati, OH).

The investigators will initially evaluate the potential benefit, risks and impact on the patient's quality of life of this modified surgical technique in 5 patients.

Expected results: The potential advantages to the patients entered into this study result from the avoidance of open or laparoscopic surgery with the related risks (bleeding, injury of organs, post operative wound infection, hernia), shorter hospital stay, reduced postoperative pain, earlier return to work, and cosmetic advantage.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo general anesthesia
* Age > 18 yrs. of age and < 85 yrs. of age
* Ability to give informed consent

Exclusion Criteria:

* Contraindicated for esophagogastroduodenoscopy (EGD)
* Contraindicated for colonoscopy
* BMI < 40
* Presence of esophageal stricture
* Altered gastric anatomy
* Intraabdominal abscess or severe inflammation
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
fistula or perforation closure possible; yes or no | day of surgery

SECONDARY OUTCOMES:
fistula stays closed after 6 months | 6 months
quality of life comparison, pre-op and after 6 months post-op | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee L Swanstrom, MD, FACS, Principal Investigator — Legacy Health System
Locations (1):
- Good Samaritan Hospital, Legacy Health System, Portland, Oregon, United States

REFERENCES:
- [Background] Sumiyama K, Gostout CJ, Rajan E, Bakken TA, Deters JL, Knipschield MA. Endoscopic full-thickness closure of large gastric perforations by use of tissue anchors. Gastrointest Endosc. 2007 Jan;65(1):134-9. doi: 10.1016/j.gie.2006.01.050. PMID 17185093
- [Background] Raju GS, Fritscher-Ravens A, Rothstein RI, Swain P, Gelrud A, Ahmed I, Gomez G, Winny M, Sonnanstine T, Bergstrom M, Park PO. Endoscopic closure of colon perforation compared to surgery in a porcine model: a randomized controlled trial (with videos). Gastrointest Endosc. 2008 Aug;68(2):324-32. doi: 10.1016/j.gie.2008.03.006. Epub 2008 Jun 17. PMID 18561931
- [Background] Sporn E, Miedema BW, Bachman SL, Astudillo JA, Loy TS, Calaluce R, Thaler K. Endoscopic colotomy closure after full thickness excision: comparison of T fastener with multiclip applier. Endoscopy. 2008 Jul;40(7):589-94. doi: 10.1055/s-2008-1077377. PMID 18609453
- [Background] Bergstrom M, Swain P, Park PO. Early clinical experience with a new flexible endoscopic suturing method for natural orifice transluminal endoscopic surgery and intraluminal endosurgery (with videos). Gastrointest Endosc. 2008 Mar;67(3):528-33. doi: 10.1016/j.gie.2007.09.049. PMID 18294516
- See also: Evaluation of an Endoscopic Suturing System for Tissue Apposition in Colonic Polypectomy — http://www.clinicaltrials.gov/ct2/show/NCT00553436